CLINICAL TRIAL: NCT05108714
Title: The Use of MicronJet600 Microneedle for Intradermal Lidocaine Injection to Ensure Local Anaesthesia During Insertion of Peripheral Venous Catheters
Brief Title: Intradermal Lidocaine Via MicronJet600 Microneedle Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: NanoPass Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.1.
Record Dates: First submitted 2021-09-21; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-09

CONDITIONS: Local Anaesthesia
Keywords: Microneedles, local anaesthesia, intradermal administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1. Left arm. (Experimental): Healthy subjects, who underwent the following intervention: intradermal injection of lidocaine hydrochloride injectable solution via MicronJet600 microneedle device at the site of antecubital fossa of the left arm, followed by the insertion of 18G catheter in a cubital vein.
  Interventions: Device: Intravenous cannulation after intradermal injection of lidocaine via MicronJet600 microneedle device (1)
- Group 1. Right arm. (Placebo Comparator): Healthy subjects, who underwent the following intervention: intradermal injection of sterile saline via MicronJet600 microneedle device at the site of antecubital fossa of the right arm, followed by the insertion of 18G catheter in a cubital vein.
  Interventions: Device: Intravenous cannulation after intradermal injection of saline via MicronJet600 microneedle device
- Group 2. Left arm. (Experimental): Healthy subjects, who underwent the following intervention: intradermal injection of lidocaine hydrochloride injectable solution via MicronJet600 microneedle device at the site of antecubital fossa of the left arm, followed by the insertion of 18G catheter in a cubital vein.
  Interventions: Device: Intravenous cannulation after intradermal injection of lidocaine via MicronJet600 microneedle device (2)
- Group 2. Right arm. (Active Comparator): Healthy subjects, who underwent the following intervention: insertion of 18G catheter in a cubital vein at the site of antecubital fossa of the right arm, without any prior intervention.
  Interventions: Procedure: Intravenous cannulation after without prior interventions

INTERVENTIONS:
Device: Intravenous cannulation after intradermal injection of lidocaine via MicronJet600 microneedle device (1) — Intradermal administration of 100 µL of lidocaine (registrational number LS001516 by Federal Service for Surveillance in Healthcare of Russian Federation) via MicronJet600 microneedle device at the site of antecubital fossa of the left arm, followed by the insertion of 18G catheter in a cubital vein immediately after the lidocaine administration.
  Arms: Group 1. Left arm.
Device: Intravenous cannulation after intradermal injection of saline via MicronJet600 microneedle device — Intradermal administration of 100 µL saline (registration number РN002134/01 by Federal Service for Surveillance in Healthcare of Russian Federation) via MicronJet600 microneedle device at the site of antecubital fossa of the right arm, followed by the insertion of 18G catheter in a cubital vein immediately after the saline administration.
  Arms: Group 1. Right arm.
Device: Intravenous cannulation after intradermal injection of lidocaine via MicronJet600 microneedle device (2) — Intradermal administration of 100 µL of lidocaine (registrational number LS001516 by Federal Service for Surveillance in Healthcare of Russian Federation) via MicronJet600 microneedle device at the site of antecubital fossa of the left arm, followed by the insertion of 18G catheter in a cubital vein immediately after the lidocaine administration.
  Arms: Group 2. Left arm.
Procedure: Intravenous cannulation after without prior interventions — insertion of 18G catheter in a cubital vein without prior interventions.
  Arms: Group 2. Right arm.

SUMMARY:
The purpose of this study is to determine efficiency and safety of injecting a micro-amount of 2% lidocaine with the commercially available microneedle device MinronJet600 (NanoPass Technologies Ltd, Israel) (registration number RZN2017/5544 by Federal Service for Surveillance in Healthcare of Russian Federation) to achieve rapid local anesthesia for peripheral venous cannulation.

DETAILED DESCRIPTION:
The trial is prospective, randomised, open-label, placebo-controlled. The start date of patient enrolment was January 29 of 2019. Simple randomization was performed to allocate subjects into two groups using the Microsoft Excel random number generator. As a result of randomisation, subjects were allocated into two groups - Group1 and Group2.

In this study, each subject from Group1 received injection of local anaesthetic into the left arm and sterile saline as a placebo into the right arm, the injections were performed with MicronJet600 and followed by the intravenous cannulation; each subject from Group2 will receive injection of local anaesthetic into the left arm, which was performed with MicronJet600 and followed by the intravenous cannulation, with no pre-treatment prior to the intravenous cannulation in case of the right arm. Pain caused by the cannulations was rated by the subjects in accordance with 100-point visual analogue scale. Safety parameters was assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Age at 18-65 years

Exclusion Criteria:

* Pregnant or lactating women
* Evidence of allergy to lidocaine
* Presence of pain of any localization and character not associated with the study or treatment with any analgesics
* Any perceptual disorders
* Neuropathies or stroke in anamnesis
* Any psychiatric disorders
* Any disorder of tissues at the site of intervention - the antecubital fossa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-17 (Actual)

PRIMARY OUTCOMES:
Pain scores, reported by the subjects due to painful stimulus by intravenous catheterisation with 18G cannula | Immediately after intravenous catheterisation with 18G cannula.
  Pain scores experienced by the subjects due to intravenous catheterisation with 18G cannula. were recorded by using a 100-point visual analogue scale.
Pain scores, reported by the subjects due to painful stimulus due to a pin-prick with a 27G needle (1) | At 15 minutes after the intradermal lidocaine injection.
  Pain scores experienced by the subjects due to a pin-prick with a 27G needle at 1, 2 and 3 centimetres from the site of intradermal lidocaine injection were recorded by using a 100-point visual analogue scale.
Pain scores, reported by the subjects due to painful stimulus due to a pin-prick with a 27G needle (2) | At 30 minutes minutes after the intradermal lidocaine injection.
  Pain scores experienced by the subjects due to a pin-prick with a 27G needle at 1, 2 and 3 centimetres from the site of intradermal lidocaine injection were recorded by using a 100-point visual analogue scale.
Pain scores, reported by the subjects due to painful stimulus due to a pin-prick with a 27G needle (3) | At 45 minutes after the intradermal lidocaine injection.
  Pain scores experienced by the subjects due to a pin-prick with a 27G needle at 1, 2 and 3 centimetres from the site of intradermal lidocaine injection were recorded by using a 100-point visual analogue scale.
Prevalence of adverse events. | 24 hours after the lidocaine injection with MicronJet600.
  Any kind of local and systemic adverse events were recorded after the lidocaine injection with MicronJet600 followed by the intravenous cannulation.

SECONDARY OUTCOMES:
Preference to receive injection of lidocaine with MicronJet600 prior to intravenous cannulation, over the cannulation without any pre-treatment. | Immediately after the intravenous catheterisation with 18G cannula.
  Preference to receive injection of lidocaine with MicronJet600 before intravenous cannulation over the cannulation without any pre-treatment in subjects of Group2. The preference was recorded with the 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Chavdar Dr Pavlov, MD, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- University Clinical Hospital №2 (I.M. Sechenov First Moscow State Medical University (Sechenov University)), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
The local ethics committee of the Sechenov University does not allow to share IPD; it is possible only upon an official request addressed to the principal investigator.

REFERENCES:
- [Derived] Rzhevskiy A, Popov A, Pavlov C, Anissimov Y, Zvyagin A, Levin Y, Kochba E. Intradermal injection of lidocaine with a microneedle device to provide rapid local anaesthesia for peripheral intravenous cannulation: A randomised open-label placebo-controlled clinical trial. PLoS One. 2022 Jan 31;17(1):e0261641. doi: 10.1371/journal.pone.0261641. eCollection 2022. PMID 35100279